CLINICAL TRIAL: NCT02154009
Title: Clinical Autonomic Disorders: A Training Protocol
Status: Terminated | Type: Observational
Why Stopped: Training protocol with no research objectives
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140122; 14-N-0122
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Posttraumatic Stress Disorder; Pseudopheochromocytoma; Healthy Volunteers; Neurocardiogenic Syncope; Postural Tachycardia Syndrome
Keywords: Autonomic Nervous System; Catecholamines; Dysautonomia; Sympathetic Cholinergic System; Sympathetic Adrenergic System
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, skin biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Volunteers will be studied for Fellows to practice and gain normative values for pupillometric function.
- Patients: Referred patients with known or suspected abnormalities of one or more components of the autonomic nervous system

SUMMARY:
Background:

- The autonomic nervous system helps control things that happen automatically in the body, like blood pressure, heart rate, and digestion. When it doesn t work properly, it s called dysautonomia. Researchers want to learn more about dysautonomias and train doctors to learn how to better diagnose them.

Objectives:

* To allow people with autonomic disorders to be evaluated.
* To help fellows in the NIH Autonomic Disorders fellowship program see a variety of diseases in their training.

Eligibility:

* People age 18 and older with dysautonomia; children over age 2 if they might benefit
* Healthy adult volunteers

Design:

* Participants will have different procedures depending on their symptoms. They will have one or more visits. They will have some but not all of the tests below.
* Participants will have a medical history and physical exam. They may be tested for problems thinking. They may complete a symptom questionnaire. They may have their temperature and blood pressure taken.
* Participants may have an intravenous line placed. A needle will guide a thin plastic tube into an arm vein.
* Participants may have blood drawn several times. They may give a urine sample.
* Participants may have an electrocardiogram.
* How much blood a participant s heart is pumping and/or how much blood is flowing through their arm may be measured. The total amount of blood in their bloodstream may be measured.
* Participants may have their ability to sweat and/or sense of smell tested.
* Breathing, bowel sounds, and/or body functions may be monitored.
* Pupil size, response to environmental temperature changes, and/or breathing may be measured.
* Participants may have a bladder ultrasound.
* Small pieces of skin may be taken for study.

DETAILED DESCRIPTION:
Objective:

This Protocol is to facilitate training of Fellows in evaluation of clinical disorders of the autonomic nervous system. The training is necessary to enable Fellows to sit for and pass the certifying examination in autonomic disorders administered by the United Council for Neurologic Subspecialties (UCNS) and to maintain UCNS accreditation of the Fellowship. A secondary objective is to include results of evaluations and testing with those from other Protocols, for future data analyses.

Study population:

Referred patients with known or suspected abnormalities of one or more components of the autonomic nervous system and healthy adult volunteers. Volunteers will be studied for Fellows to practice and gain normative values for pupillometric function.

Design:

Clinical physiologic, neuropharmacologic, and neurochemical testing will be performed during outpatient clinic visits or during inpatient admissions, depending on the individual testing schedule. Inpatient testing may be done in conjunction with other Protocols (e.g., 03-N-0004). Most of the testing under this Protocol can be completed in a single outpatient visit over the course of a workday. Testing procedures under this Protocol will be performed as needed for adequate Fellow training. In addition to autonomic medical history and physical examination, clinical testing procedures may include (A) monitoring of hemodynamics, sweating, and other physiologic parameters associated with the Valsalva maneuver, orthostasis, or external temperature manipulation; (B) venous blood sampling for assays of levels of catecholamines and related neurochemicals; (C) administration of autonomic test drugs; (D) skin biopsies; (E) blood volume measurement; (F) pupillometry; (G) gastrointestinal phonography; (H) urinary bladder ultrasound; and (I) neurobehavioral rating scales.

Outcome measures:

The main outcome measure is competency in clinical and laboratory evaluation of autonomic disorders, based on assessment of the Fellow by the Principal Investigator at approximately 6-month intervals. A secondary outcome measure is results obtained under this Protocol, which may be analyzed and reported as research data along with data from other Protocols.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENTS:

Patients may be included if they are at least 18 years old and are known or suspected to have failure of one or more components of the autonomic nervous system, small fiber neuropathy, inherited dysautonomia, orthostatic intolerance, neurocardiogenic syncope, status post endoscopic thoracic sympathectomy, or disorders of catecholamine synthesis or fate.

Children greater than two years old may be enrolled in this Protocol if they might personally benefit from the tests in the Protocol through the establishment of a diagnosis.

EXCLUSION CRITERIA - PATIENTS:

There are no exclusion criteria for the study as a whole.

INCLUSION CRITERIA - HEALTHY VOLUNTEERS:

Healthy adult Volunteers (at least 18 years old) may be included, pending normal or medically insignificant results of history and physical examination. A repeat history and physical examination is required if more than 6 months have gone by from a previous workup.

EXCLUSION CRITERIA - HEALTHY VOLUNTEERS:

A candidate Healthy Volunteer will be excluded if the person has any of the following: symptoms of autonomic dysfunction, including lightheadedness, fainting, abnormalities of sweating, frequent nausea, vomiting, constipation, or diarrhea, or urinary frequency or retention. If the Volunteer has a condition requiring medication that in the judgment of the Investigators will affect results of the pupillometric tests under this Protocol, the Volunteer may be included for training purposes.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Referred patients with known or suspected abnormalities of one or more components of the autonomic nervous system and healthy adult volunteers. Volunteers will be studied for Fellows to practice and gain normative values for pupillometric function.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Successful completion of the Clinical Fellowship in autonomic disorders | approximately 6-month intervals.
  Competency in clinical and laboratory evaluation of autonomic disorders, based on assessment of the Fellow by the Principal Investigator at approximately 6-month intervals

SECONDARY OUTCOMES:
Clinical samples and data from evaluation of patients with known or suspected autonomic disorders | Initial Visit
  Analysis of clinical samples and data from evaluation of patients with known or suspected autonomic disorders reported as research data along with data from other Protocols.

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-N-0122.html